CLINICAL TRIAL: NCT05202691
Title: Comparison of the Effects of Physical Therapy With and Without Magnetic Field Therapy in People With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ComplutenseHolystic
Record Dates: First submitted 2021-12-09; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Low Back Pain
Keywords: low back pain; physical therapy; rehabilitation; magnetic field therapy
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities; Magnetic Field Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial evaluating clinical effects in people with low back pain who are divided into 2 groups of treatment, where the interventions are conducted in 3 sessions provided during 3 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To participants: the intervention applied to both groups is the same Physical Therapy Treatment protocol and the use of the same magnetic field therapy device during the same time (for the sham group: the device is disconnected and the sound is simulated with a recording).
  The investigator assessing the outcomes is blinded to the group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Physical Therapy+Magnetic Field Therapy) (Experimental): Physical Therapy Protocol plus Magnetic Field Therapy
  A protocol of physical therapy treatment including:
  * Manual therapy techniques for inhibition of piriformis, quadratus lumbaris, and paravertebral muscles in prone position and bilaterally.
  * 2 functional techniques applied to the sacrum in prone position.
  * A myofascial release of ligaments inserted to the sacrum in prone position and bilaterally.
  * Manual therapy technique for inhibition of psoas-iliacus muscle in supine position and bilaterally.
  * Stretching techniques of piriformis, gluteal and paravertebral muscles in supine position and bilaterally.
  * Active gluteus maximus contraction in supine position bilaterally.
  To this protocol, a 15 minutes of Magnetic Field Therapy using the Zimmer EmfieldPro device (Zimmer MedizinSysteme, Germany) applied to the lumbosacral region in prone position is added.
  Interventions: Other: Group 1 (Physical Therapy+Magnetic Field Therapy)
- Group 2 (Physical Therapy) (Active Comparator): Physical Therapy Protocol alone:
  The same Physical Therapy Treatment protocol with a sham magnetic intervention applying in the same region with a disconnected Zimmer EmfieldPro device (Zimmer MedizinSysteme, Germany) during 15 minutes.
  Interventions: Other: Group 2 (Physical Therapy)

INTERVENTIONS:
Other: Group 1 (Physical Therapy+Magnetic Field Therapy) — A Physical Therapy Protocol (including manual therapy, stretching and exercise for low back pain) adding a Magnetic Field Therapy using the Zimmer EmfieldPro device (Zimmer MedizinSysteme, Germany)
  Other Names: physical therapy and magnetic field therapy for low back pain
  Arms: Group 1 (Physical Therapy+Magnetic Field Therapy)
Other: Group 2 (Physical Therapy) — A Physical Therapy Protocol (including manual therapy, stretching and exercise for low back pain)
  Other Names: physical therapy for low back pain
  Arms: Group 2 (Physical Therapy)

SUMMARY:
A randomized and controlled trial to people with low back pain who are divided into 2 groups of treatment: 1- people treated with a protocol of physical therapy techniques without magnetic field therapy; 2- people treated with the same protocol of physical therapy techniques adding a magnetic stimulation treatment. The interventions are conducted in 3 sessions provided during 3 weeks.The lumbar pain and disability are assessed before and after the intervention, and lumbar flexion and extension pain are assessed before and after each session in all the participants.

DETAILED DESCRIPTION:
This study is a randomized controlled trial evaluating clinical effects of a protocol of Physical Therapy Treatment (PTT), via manual therapy and active mobilization, adding or not a magnetic field therapy in people with non-specific low back pain lasting at least 6 weeks. Participants were randomized to receive either a PTT protocol including a magnetic stimulation treatment or the same PTT protocol with a sham magnetic intervention. The interventions are conducted in 3 sessions provided during 3 weeks.

Intervention:

A description of the 2 groups of treatment:

1. - Experimental group 1: a protocol of physical therapy treatment including:

   * Manual therapy techniques for inhibition of piriformis, quadratus lumbar, and paravertebral muscles in prone position and bilaterally.
   * 2 functional techniques applied to the sacrum in prone position.
   * A myofascial release of ligaments inserted to the sacrum in prone position and bilaterally.
   * Manual therapy technique for inhibition of psoas-iliacus muscle in supine position and bilaterally.
   * Stretching techniques of piriformis, gluteal and paravertebral muscles in supine position and bilaterally.
   * Active gluteus maximus contraction in supine position bilaterally.

   To this protocol, a 15 minutes of magnetic field therapy treatment applied to the lumbosacral region in prone position is added.
2. - Experimental group 2: the same Physical Therapy Treatment protocol with a sham magnetic intervention applying in the same region with a disconnected device during 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were individuals aged between 18 and 65 years with a diagnosis of non-specific low back pain, with or without lower limb irradiation, lasting at least 6 weeks.

Exclusion Criteria:

* Pregnancy, spinal tumor or infection, diabetes, spinal fracture or previous spine surgery.
* Patients with a history of rehabilitation treatment for back pain within the preceding month
* Unstable medical disorder not controlled by standard treatment and those with a cardiac pacemaker or using any other electrical devices or prosthesis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Lumbar pain change with the Pain Detect Questionnaire | Change from Baseline Lumbar pain at 4 weeks.
  lumbar pain at this moment and in the last 4 weeks evaluated with the Pain Detect Questionnaire. The Questionnaire has a maximum score of 35 and a minimum score of 0. Lower scores mean a better outcome.
Disability Questionnaire 1 change | Change from Baseline degree of diability at 4 weeks.
  Disability Questionnaire assessed with the Roland-Morris Questionnaire. The Questionnaire has a maximum score of 24 and a minimum score of 0. Lower scores mean a better outcome.
Disability Questionnaire 2 change | Change from Baseline degree of diability at 4 weeks.
  Disability Questionnaire 2 assessed with the Oswestry Disability Index. The Oswestry Disability Index is scored from 0 (absence of disability) to 100 (maximum disability). This questionnaire has 10 multiple-choice questions, each of which may be scored between 0 (no disability) and 5 (maximum disability). Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Lumbar flexion Numerical Rating Scale | 4 weeks (immediately before and after each of the sessions)
  Lumbar flexion evaluated with a Numerical Rating Scale. The minimum value is 0 and the maximum value is 10. Lower scores mean a better outcome.
Lumbar extension Numerical Rating Scale | 4 weeks (immediately before and after each of the sessions)
  Lumbar extension evaluated with a Numerical Rating Scale. The minimum value is 0 and the maximum value is 10. Lower scores mean a better outcome.
Finger to Floor test | 4 weeks (immediately before and after each of the sessions)
  Lumbar mobility evaluated with the finger-to-floor test, assessed before and after each session in all the participants. The minimum value is 0 centimeters and the maximum value depending the flexibility os each participant and the distance, in centimeters between fingers anthe floor. Lower distance in centimeters means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Isidro Fernández-López, Dr., Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markov MS. Magnetic field therapy: a review. Electromagn Biol Med. 2007;26(1):1-23. doi: 10.1080/15368370600925342. PMID 17454079
- [Background] Daish C, Blanchard R, Fox K, Pivonka P, Pirogova E. The Application of Pulsed Electromagnetic Fields (PEMFs) for Bone Fracture Repair: Past and Perspective Findings. Ann Biomed Eng. 2018 Apr;46(4):525-542. doi: 10.1007/s10439-018-1982-1. Epub 2018 Jan 22. PMID 29356996
- [Background] Hu H, Yang W, Zeng Q, Chen W, Zhu Y, Liu W, Wang S, Wang B, Shao Z, Zhang Y. Promising application of Pulsed Electromagnetic Fields (PEMFs) in musculoskeletal disorders. Biomed Pharmacother. 2020 Nov;131:110767. doi: 10.1016/j.biopha.2020.110767. Epub 2020 Sep 23. PMID 33152929